CLINICAL TRIAL: NCT01352195
Title: Extended Self-Help for Smoking Cessation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MCC-15724
Record Dates: First submitted 2011-05-10; First posted 2011-05-11 (Estimated); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: Smoking Cessation
Keywords: Forever Free
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Usual Care (UC) (Active Comparator): This condition will comprise a single, high quality booklet that is currently in dissemination: NCI's Clearing the Air (NCI, 2003).
  Interventions: Behavioral: Forever Free Booklets
- Standard Repeated Mailings (Stand-RM) (Active Comparator): Stand-RM will be the same 8 Forever Free booklets (edited for cessation) distributed over 12 months as in our preliminary studies.
  Interventions: Behavioral: Forever Free Booklets
- Intensive Repeated Mailings (Inten-RM) (Active Comparator): Inten-RM will add two additional booklets to extend the intervention out to 18 months, plus additional monthly contacts.
  Interventions: Behavioral: Forever Free Booklets

INTERVENTIONS:
Behavioral: Forever Free Booklets — Randomized 3-arm design, with 660 smokers recruited into each condition. Assessments will occur at six-month intervals, through 30 months.

SUMMARY:
The primary purpose of this study is smoking cessation. The investigators are conducting a research study to learn how well the information from the program helps participants to quit smoking and remain smoke-free.

DETAILED DESCRIPTION:
The investigators propose a randomized 3-arm design, with 660 smokers recruited into each condition. The three conditions will include: (1) Usual care (UC), which will comprise a single smoking cessation booklet developed by NCI; (2) Standard Repeated Mailings (Stand-RM), which will be the same 8 Forever Free booklets (edited for cessation) distributed over 12 months as in our preliminary studies; and (3) Intensive Repeated Mailings (Inten-RM), which will add two additional booklets to extend the intervention out to 18 months, plus additional monthly contacts. Assessments will occur at six-month intervals, through 30 months. An overview of the design is depicted in Table 4, which will be referenced throughout the remainder of this proposal.

ELIGIBILITY:
Participants:

* Planned Participants: 1980 daily smokers (for a final sample of at least 1584 after attrition), recruited via multimedia advertisements (daily and weekly newspapers, radio, cable television, public transit ads, etc.), public service announcements, and direct community engagement.

Inclusion Criteria:

* smoking at least five cigarette per day over the past year
* not currently enrolled in a face-to-face smoking cessation program
* able to speak and read English
* desire to quit smoking, as indicated by a score of at least 5 ("Think I should quit, but not quite ready") on the Contemplation Ladder (Biener & Abrams, 1991)

Exclusion Criteria:

* number of participants from the same street address limited to 1
* no more than 2 referrals per participant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2124 (Actual)
Dates: Start 2009-01-23 (Actual); Primary Completion 2014-02-18 (Actual); Study Completion 2014-08-27 (Actual)

PRIMARY OUTCOMES:
7-Day Point-Prevalence Abstinence at Each Follow-up Point | 30 months per participant
  Time will be measured in months from the start of condition. Potential confounding variables (e.g., group differences in demographic, smoking history, or pharmacotherapy use) will be adjusted for in the model. Pair-wise condition and time interval comparisons will be tested using the generalized score statistics from generalized estimating equations (GEE) models by utilizing the contrast statements.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Brandon, Ph.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

REFERENCES:
- [Derived] Brandon TH, Simmons VN, Sutton SK, Unrod M, Harrell PT, Meade CD, Craig BM, Lee JH, Meltzer LR. Extended Self-Help for Smoking Cessation: A Randomized Controlled Trial. Am J Prev Med. 2016 Jul;51(1):54-62. doi: 10.1016/j.amepre.2015.12.016. Epub 2016 Feb 8. PMID 26868284